CLINICAL TRIAL: NCT00531362
Title: Enteric Coating as a Factor in Aspirin Resistance
Status: Completed | Type: Observational
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: Irish Heart Foundation (Other)
Responsible Party: Dermot Cox, Royal College of Surgeons in Ireland
Other Study IDs: RCSI1
Record Dates: First submitted 2007-09-17; First posted 2007-09-18 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-09

CONDITIONS: Cardiovascular Disease
Keywords: Atherosclerosis; Aspirin; Resistance,; Acute coronary syndromes
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples will be collected and stored for later analysis
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients: All patients (acute or stable) presenting to a cardiovascular clinic and on aspirin.
  Interventions: Drug: Plain aspirin

INTERVENTIONS:
Drug: Plain aspirin — Plain aspirin 75 mg or 150 mg

SUMMARY:
Aspirin is an essential drug for the treatment of cardiovascular disease. The standard dose is 75mg per day (much lower than that for inflammation or fever). One of the side-effects of aspirin is a gastric ulcer which can be fatal. To prevent this it is common to use enteric-coated aspirin. This passes through the stomach intact and dissolves in the intestines. This prevents high levels of drug forming in the stomach reducing ulcer formation. Recently there is evidence of high levels of aspirin resistance, ie, patients who appear not to achieve the maximum benefit from aspirin. Clinical studies have shown a significant increase in mortality among these patients.

A recent study that we performed showed that enteric-coated aspirin is not as effective as plain aspirin. This was especially noticeable in heavier volunteers. In fact it appeared that enteric-coated aspirin only delivers 50mg aspirin instead of the full 75 mg. For volunteers resistant to enteric-coated aspirin simply switching them to plain aspirin solved the problem.

We propose to recruit patients on 75 mg enteric aspirin and test them for evidence of poor response to aspirin. Poor responders will then be given 75mg plain aspirin and tested for their response. Those that fail to respond will then receive 150 mg aspirin. If the results of the healthy volunteer study are replicated this would provide a very cheap and effective solution to a serious problem.

DETAILED DESCRIPTION:
In a recent study we have shown clear evidence for pharmacokinetic aspirin resistance in healthy volunteers due to poor bioavailability of enteric-coated aspirin. However, it is necessary to confirm that pharmacokinetic resistance is an important factor in aspirin resistance in a patient population as well. To achieve this we will compare the response of patients to enteric-coated aspirin and plain aspirin in an open-labeled cross-over study in patients undergoing treatment with enteric-coated aspirin.

Patient population: Patients will be recruited from Dr. David Foley's clinic in Beaumont Hospital. All patients who have been prescribed enteric-coated aspirin (75 mg, any brand) will be considered eligible for enrollment providing they are competent to give informed consent. Patients of any diagnosis, any age and those on other medication will be considered eligible. Patients who are likely to stop aspirin therapy within a few weeks due to planned surgery or who are showing signs of adverse effects to aspirin will be excluded. Patients already enrolled in a clinical study will also be excluded.

Study design: After obtaining informed consent an appointment will be made with a patient to return to give a blood sample (ideally 1-2 weeks). The patient will be reminded of the importance of compliance and asked to keep a diary of aspirin use. On the scheduled visit a blood sample will be taken and the patient will be advised to keep taking their aspirin and that they would be advised of the outcome of the test within a week.

After the platelet function assessment those patients with adequate inhibition of platelet function will be informed that their aspirin dose is fine, reminded of the importance of compliance and their role in the study terminated. Patients who do not meet the target level of inhibition will be asked to return to the hospital where they will be switched to plain aspirin. They will be asked to return after two weeks for a further visit. Platelet function will then be assessed again. If the target inhibition is achieved they will be terminated from the study and with the agreement of their physician they will be switched to plain aspirin for future use. Those patients who do not achieve the target inhibition will be switched to 150 mg plain aspirin daily. A final escalation to 300 mg will used if necessary.

Platelet function tests Serum thromboxane. The gold-standard test of aspirin effects will be serum thromboxane production as determined by ELISA. A 5ml blood sample will be collected into a serum tube and incubated at 37ºC for 30 mins. The tube will then be centrifuged and the serum removed and frozen at -20ºC until analysed. In a previous study the baseline serum thromboxane levels in healthy volunteers was 276±99 ng/ml (±SD; n=142) and thus 95% inhibition would represent 13 ng/ml. We have previously shown that a serum thromboxane value of 2.2 ng/ml is a more effective marker of platelet function. This test will be unaffected by other medications except for anti-coagulants such as warfarin.

Arachidonic acid-induced aggregation. A second test to measure the effectiveness of aspirin is arachidonic acid-induced aggregation. Blood will be collected into sodium citrate and centrifuged to generate platelet-rich plasma. Arachidonic acid will be

Experimental design (continued)

added to PRP and stirred in a platelet aggregometer. In healthy volunteers plain aspirin reduced the aggregation response to 4% aggregation.

Supernatant thromboxane. We have recently developed a novel assay that is extremely sensitive to inhibition by aspirin. This is in effect a combination of the two assays described above. The supernatant from the arachidonic acid-induced aggregation experiment will be collected and frozen at -20ºC. The thromboxane levels in these samples will be determined by ELISA.

Verify Now (aspirin): Point-of-care assays are very useful for diagnosing aspirin resistance. It allows instantaneous feedback for the doctor and allows remedial action to be taken immediately. One of the more effective point-of-care devices is the Ultegra Verify Now device from Accumetrics. This is a cartridge-based system that monitors aggregation in response to arachidonic acid in whole blood. A small aliquot of blood will be tested for aspirin resistance using the Verify Now assay.

Study outcome.

1. This study will provide an estimate of the incidence of incomplete inhibition of COX in patients on enteric coated aspirin. We plan on recruiting 50 patients with <95% inhibition which will provide a margin of error of 15% on the estimate.
2. We will determine if enteric-coating of aspirin is responsible for this incomplete inhibition.
3. We will determine if patients with incomplete inhibition of COX on plain aspirin can benefit from an increased dose of aspirin.
4. We will obtain data on the sensitivity and reliability of various aspirin response assays.

Benefits of the research. Cardiovascular disease is still the major cause of death in Ireland today. Treatment with low-dose aspirin is a key strategy in preventing further cardiovascular events. Recently enteric-coated aspirin preparations have become standard despite the paucity of information on their bioequivalence to plain aspirin. The poorly defined phenomenon of aspirin resistance has been shown to adversely impact on the benefits of aspirin therapy and this has been associated with the use of enteric-coated aspirin. This study will allow us to quantify the extent of aspirin non-response in patients on enteric-coated aspirin and confirm if the use of plain aspirin will overcome this resistance. This will provide a very cost-effective solution to a major problem in cardiovascular disease treatment strategies.

ELIGIBILITY:
Inclusion Criteria:

* Stable or unstable coronary artery disease
* On aspirin

Exclusion Criteria:

* Inability to give informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients attending the cardiac outpatients clinic or the cat lab of Beaumont hospital, Dublin, Ireland
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2007-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dermot Cox, PhD, Principal Investigator — Royal College of Surgeons
Locations (1):
- Beaumont Hospital, Dublin, Ireland

REFERENCES:
- [Background] Cox D, Maree AO, Dooley M, Conroy R, Byrne MF, Fitzgerald DJ. Effect of enteric coating on antiplatelet activity of low-dose aspirin in healthy volunteers. Stroke. 2006 Aug;37(8):2153-8. doi: 10.1161/01.STR.0000231683.43347.ec. Epub 2006 Jun 22. PMID 16794200
- See also: Irish Heart Foundation, study sponsor website — http://www.irishheart.ie/